CLINICAL TRIAL: NCT05209347
Title: Custom Dynamic Orthoses to Reduce Articular Contact Stress
Acronym: PRMRP FPA CT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study related activities were delayed and effort was instead focused on recruitment and testing for the iterative design study (NCT04562896).
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jason Wilken, Director of Collaborative Research and Development, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 202112331; CDMRP-PR172087 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2023-12

CONDITIONS: Ankle Fractures; Post-traumatic Osteoarthritis; Osteoarthritis Ankle
Keywords: Carbon Fiber; Gait Analysis; Ankle Foot Orthosis; Arthritis; Biomechanics; Ankle; Adult
MeSH Terms: conditions — Ankle Fractures; Arthritis

STUDY DESIGN:
Intervention Model Description: All participants will be cast and fit with two CDOs. Each CDO will be labeled as CDO-A or CDO-B. Participants will be randomly assigned to one of two CDO testing sequences (AB, BA) to prevent testing order from influencing study results.
Who Masked: Participant
Masking Description: Participants will be blinded to the different CDO designs and will only be introduced to each device as CDO-A or CDO-B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- NoCDO (No Intervention): Participants will be evaluated without a CDO
- CDO-A (Experimental): The first study CDO will be designated CDO-A
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- CDO-B (Experimental): The second study CDO will be designated CDO-B
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)

INTERVENTIONS:
Device: Carbon Fiber Custom Dynamic Orthosis (CDO) — The carbon fiber custom dynamic orthosis will consist of a semi-rigid foot plate, a posterior carbon fiber strut, and a proximal cuff below the knee.
  Other Names: Ankle Foot Orthosis (AFO)
  Arms: CDO-A; CDO-B

SUMMARY:
The proposed study evaluates the effect of carbon fiber brace design on forces across the ankle. Research suggests that ankle arthritis develops following ankle fracture due, in part, to elevated forces on the cartilage. It is expected that carbon fiber braces can reduce forces in the ankle joint thereby reducing the risk of developing arthritis following injury. In this study, carbon fiber braces will be tested to determine how they influence the forces acting on the ankle cartilage. The proposed study will provide evidence that can be used by clinicians and researchers to design carbon fiber braces to effectively reduce forces on ankle cartilage.

DETAILED DESCRIPTION:
The primary purpose of this line of research is to investigate the effects of carbon fiber custom dynamic orthosis (CDO) use on forces and contact stress at the ankle, with the goal of reducing the development of post traumatic osteoarthritis (PTOA). Research suggests that PTO develops, in part, due to increased ankle contact stress following fracture. It is expected that reducing articular contact stress has the potential to delay or prevent PTOA development. CDOs have been shown to significantly improve function after extremity injury, and show promise for offloading the injured ankle joint after severe lower extremity injuries. Therefore, the proposed effort is designed to evaluate CDOs effects on forces and articular contact stress at the ankle.

Adult participants who have sustained a traumatic ankle fracture of the tibial pilon will be evaluated while wearing two CDOs, with a primary dependent measure of ankle joint contact stress. Following consent and enrollment weight bearing computerized tomography (CT) images will be collected and used to determine the geometry of the joint, and the articular contact stress using discrete element analysis.

Participants will be cast and fit for two CDOs. Participants will be blinded to the design variation of each device and will only know them as CDO-A or CDO-B. Testing will be completed under 3 conditions: No-CDO, CDO-A, CDO-B, with each bracing condition (A/B) representing a different CDO. Physical performance measures will incorporate tests of agility, speed, and lower limb power to ensure that the CDOs do not negatively affect physical function. Questionnaires will be used to evaluate participants' current and desired activity level, pain with and without using a CDO, satisfaction with the study CDOs, perception of comfort and smoothness between CDOs, and preference between CDOs. Semi-structured interviews will be completed to fully capture the participant's perspective with each study CDO. Lower limb forces and motion will be assessed using a computerized motion capture system and force plates embedded in the floor. Forces between the foot and CDO footplate will be measured using force sensing insoles, and muscle activity data will be collected using wireless surface electromyography sensors. Each CDO will be mechanically tested, and participant demographic and anthropometric data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Sustained unilateral fracture of the tibial pilon
* The fracture has completely healed
* Ability to walk 50 feet without use of an assistive device (cane, crutch, etc.)
* Ability to walk at a slow to moderate pace
* Shoe size between women's 8 and 13.5 or men's 6.5 and 12
* Ability to read and write in English and provide written informed consent
* Individuals with elevated contact stress according to model generated using standing CT images (will be answered after completing visit one)

Exclusion Criteria:

* Pain > 6/10 while walking
* Increase in pain during testing of 3/10 or greater
* Neurologic, musculoskeletal (including bilateral fractures) or other condition limiting function of the contralateral extremity
* Medical or psychological condition that would preclude functional testing (ex. moderate or severe brain injury, stroke, heart disease)
* Wounds to the calf that would prevent CDO fitting
* Fractures secondary to neuropathy or severe osteopenia
* Classification as non-ambulatory
* Previous fractures near the tibial pilon on the involved limb
* Surgery on involved limb anticipated in the next 6 months
* Requirement of a knee stabilizing device (i.e. KAFO, KO…) to perform daily activities
* Visual or hearing impairments that limit walking ability or limit the ability to comply with instructions given during testing
* BMI greater than 40
* Pregnancy- Per participant self-report. Due to the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes, participants will be withdrawn from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Joint Contact Stress Exposure (Model estimated) | Baseline
  Joint contact stress exposure (MPA-s/gait cycle) will be estimated using a participant specific musculoskeletal model.
Peak Plantar Force (total foot) | Baseline
  Plantar forces (N) will be measured across the forefoot (100% of sensor) as participants walk without a CDO and with each CDO.
Plantar Force Impulse (total foot) | Baseline
  Plantar force impulse (Ns) across the forefoot (100% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Peak Plantar Force (forefoot) | Baseline
  Plantar forces (N) will be measured across the forefoot (distal 40% of sensor) as participants walk without a CDO and with each CDO.
Plantar Force Impulse (forefoot) | Baseline
  Plantar force impulse (Ns) across the forefoot (distal 40% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Peak Plantar Force (midfoot) | Baseline
  Plantar forces (N) will be measured across the forefoot (middle 30% of sensor) as participants walk without a CDO and with each CDO.
Plantar Force Impulse (midfoot) | Baseline
  Plantar force impulse (Ns) across the forefoot (middle 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Peak Plantar Force (hindfoot) | Baseline
  Plantar forces (N) will be measured across the forefoot (proximal 30% of sensor) as participants walk without a CDO and with each CDO.
Plantar Force Impulse (hindfoot) | Baseline
  Plantar force impulse (Ns) across the forefoot (proximal 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Numerical Pain Rating Scale | Baseline
  Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable.
Participant Device Preference | Baseline
  The participant will rank order their preference for their standard of care device (if applicable), NoCDO, CDO-A, CDO-B on a questionnaire.

SECONDARY OUTCOMES:
Four Square Step Test (4SST) | Baseline
  The 4SST (s) is a standardized timed test of balance and agility.
Sit to Stand 5 Times (STS5) | Baseline
  STS5 (s) is a well-established timed measure of lower limb muscle strength and power. Participants are instructed to stand up and sit down 5 times as fast as possible.
Ankle Range of Motion | Baseline
  Ankle range of motion (degrees) during gait.
Peak Ankle Moment | Baseline
  Peak ankle moment (Nm/kg) during gait.
Peak Ankle Power | Baseline
  Peak ankle power (W/kg) during gait.
The Orthotics Prosthetics Users' Survey (OPUS) | Baseline
  Satisfaction with device will be assessed using the Orthotics Prosthetics Users' Survey Satisfaction With Device Score (11-55). Lower scores indicate a better outcome.
Modified Socket Comfort Score (Comfort) | Baseline
  Comfort scores range from 0 = most uncomfortable to 10 = most comfortable.
Modified Socket Comfort Score (Smoothness) | Baseline
  Smoothness scores range from 0 = least smooth to 10 = most smooth.

OTHER OUTCOMES:
Semi-Structured Interview | Baseline
  Semi-structured interviews will also be used to fully capture the patients' perspectives, experience, and opinions associated with the device options they experienced as part of the study.
Center of pressure velocity timing | Baseline
  Timing of peak center of pressure velocity (percent stance) during gait.
Center of pressure velocity magnitude | Baseline
  Magnitude of peak center of pressure velocity (m/s) during gait.
Soleus Muscle Activity (Electromyography) | Baseline
  Electromyography (EMG, % Maximum) of the soleus during gait.
Tibialis Anterior Muscle Activity (Electromyography) | Baseline
  Electromyography (EMG, % Maximum) of theTibialis Anterior during gait.
Medial Gastrocnemius Muscle Activity (Electromyography) | Baseline
  Electromyography (EMG, % Maximum) of the Medial Gastrocnemius during gait.
Rectus Femoris Muscle Activity (Electromyography) | Baseline
  Electromyography (EMG, % Maximum) of the Rectus Femoris during gait.
Vastus Medialis Muscle Activity (Electromyography) | Baseline
  Electromyography (EMG, % Maximum) of the Vastus Medialis during gait.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No